CLINICAL TRIAL: NCT02943681
Title: Boosting the Beneficial Non-specific Effects of Live Attenuated Vaccines: A Randomized Controlled Trial (RCT) of a Second Dose of Measles Vaccine (MV) in the Second Year of Life
Brief Title: A Second Dose of Measles Vaccine (MV) in the Second Year of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandim Health Project (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MV18Months
Record Dates: First submitted 2016-10-13; First posted 2016-10-25 (Estimated); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Child Mortality; Child Morbidity
MeSH Terms: interventions — Measles Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Measles vaccine (Experimental): Measles vaccine, 1 dose of 0.5 ml
  Interventions: Biological: Measles vaccine
- Control (No Intervention): Nothing

INTERVENTIONS:
Biological: Measles vaccine
  Arms: Measles vaccine

SUMMARY:
This study evaluates the non-specific effects on child mortality and morbidity of a second dose of measles in the second year of life. Half of the study participants will receive a second dose of measles vaccine at 18 months of age while the other half will receive a second dose of measles by 4 years of age or at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Children need to have received the third dose of inactivated vaccines (Penta, PCV13 and IPV) before measles vaccination.

Exclusion Criteria:

* Having severe malformations that impairs their health
* Having received a second dose of measles vaccine
* Severely ill (requiring hospitalization) upon clinical examination

Ages: 18 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3812 (Actual)
Dates: Start 2016-10; Primary Completion 2020-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 months
  Mortality registered monthly by Health and Demographic Surveillance System fieldworkers. Mortality will be combined with hospital admissions in the analysis to form the outcome severe morbidity. This will be examined overall and by sex
Hospital admissions | 30 months
  Hospital admissions registered daily at the national hospital. Hospital admissions will be combined with mortality in the analysis to form the outcome severe morbidity. This will be examined overall and by sex

SECONDARY OUTCOMES:
Hospital admission by cause | 30 months
  Causes of hospital admissions registered daily at the national hospital. These will be examined overall and by sex
Consultations | 30 months
  Consultations registered daily at the local health centers and the national hospital. These will be examined overall and by sex

CONTACTS AND LOCATIONS:
Locations (1):
- Bandim Health Project, Apartado 861, Bissau, Guinea-Bissau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berendsen MLT, Silva I, Bale C, Nielsen S, Hvidt S, Martins CL, Benn CS, Aaby P. The Effect of a Second Dose of Measles Vaccine at 18 Months of Age on Nonaccidental Deaths and Hospital Admissions in Guinea-Bissau: Interim Analysis of a Randomized Controlled Trial. Clin Infect Dis. 2022 Oct 12;75(8):1370-1378. doi: 10.1093/cid/ciac155. PMID 35218356